CLINICAL TRIAL: NCT07188311
Title: A Single-arm, Open-label, Multicenter Phase II Clinical Study of Pucotenlimab Combined With Lenvatinib and Chemotherapy in the Treatment of Advanced, Relapsed/Refractory Hepatoblastoma in Children
Brief Title: Pucotenlimab Combined With Lenvatinib and Chemotherapy in the Treatment of Advanced, Relapsed/Refractory Hepatoblastoma in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Chief of Department of pediatric oncology, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2025-101-02
Record Dates: First submitted 2025-08-26; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hepatoblastoma; Pediatric Cancer
MeSH Terms: conditions — Hepatoblastoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pucotenlimab plus a fixed regimen（Lenvatinib and Irinotecan) (Experimental)
  Interventions: Drug: Pucotenlimab ,Lenvatinib

INTERVENTIONS:
Drug: Pucotenlimab ,Lenvatinib — A total of 24 cases are planned to be enrolled. All subjects will receive Pucotenlimab (3mg/kg, on Day 1, with a maximum dose not exceeding 200mg) once every 3 weeks (Q3W), in combination with Lenvatinib and Irinotecan. The chemotherapy regimen is fixed: Lenvatinib capsules 7mg/m2 (maximum 12mg) orally from Day 1 to 21 and Irinotecan 50mg/m2 from Day 1 to 5. Chemotherapy will be administered for 2 to 4 cycles, once every 3 weeks (Q3W).

SUMMARY:
This study is a single-cohort study. Pediatric patients with advanced, relapsed/refractory hepatoblastoma who have previously failed first-line or higher systemic therapy will receive 2 cycles of treatment with sintilimab combined with lenvatinib and chemotherapy (irinotecan). Patients may discontinue treatment due to disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or other reasons specified in the protocol, whichever occurs first.

* Dose setting:
* Sintilimab: The recommended dose is 3 mg/kg (maximum dose not exceeding 200 mg per administration), administered by intravenous infusion (60±15 minutes) once daily on Day 1.
* Lenvatinib: 7 mg/m² (maximum 12 mg), taken orally once daily on Days 1-21.
* Chemotherapy (irinotecan hydrochloride injection):
* Irinotecan hydrochloride injection: 50 mg/m², administered by intravenous infusion once daily on Days 1-5.
* Each 3 weeks constitutes one cycle. For patients who discontinue the study drug without radiological progression, follow-up and tumor assessment will continue until progressive disease (PD) occurs, new anti-tumor therapy is initiated, or death.
* Tumor tissues and peripheral blood of patients will be collected for relevant tests.

ELIGIBILITY:
Voluntarily enroll in the study and sign a written informed consent form; Aged 2-18 years, with no gender restrictions; Patients with histologically or cytologically confirmed locally advanced or metastatic hepatoblastoma who have received at least 1 line of systemic therapy. Participants must have experienced disease progression after previous treatment, or have relapsed or refractory disease (failure to achieve complete remission or partial remission after at least 2 courses of first-line treatment); According to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1), there is at least one radiologically measurable lesion. Lesions within the field of previous radiotherapy can be considered measurable if progression is confirmed; or there is "non-measurable disease" associated with elevated alpha-fetoprotein.

Within 3 days before the start of study treatment, the Karnofsky Performance Status score (for participants ≥16 years old) or Lansky Performance Status score (for participants <16 years old) is at least 50; Expected survival time ≥3 months; Participants with known brain metastases are eligible if they have completed primary brain treatment (such as whole-brain radiotherapy, stereotactic radiosurgery, or complete surgical resection), remain clinically stable, asymptomatic, and have discontinued steroids for at least 28 days before starting study treatment.

Archival tumor tissue or newly obtained biopsy specimens must be available for biomarker analysis before the first dose of the study drug. In cases where archival tissue cannot be provided, tumor patients who cannot obtain biopsy specimens may be enrolled without biopsy after consultation and approval by the sponsor.

Female patients of childbearing potential (i.e., not postmenopausal or not surgically sterilized) must have a negative serum pregnancy test result within 7 days before administration of the study drug; Female or male patients of childbearing potential must use reliable contraceptive measures during the administration of the study drug and within 60 days after the last dose;

Normal function of major organs, meeting the following criteria:

Routine blood test:

1. Absolute Neutrophil Count (ANC) ≥1.5×10⁹/L;
2. Platelet count ≥100×10⁹/L;

   Blood biochemistry test:
3. Total bilirubin ≤1.5×Upper Limit of Normal (ULN);
4. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5×ULN (for participants with liver metastases, ALT or AST ≤5×ULN is allowed);
5. Creatinine ≤1.5×ULN;

   Coagulation function:
6. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5×ULN;
7. Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN;
8. Myocardial enzyme profile within the normal range (isolated laboratory abnormalities deemed clinically insignificant by the investigator are allowed for enrollment).

Exclusion Criteria Received chemotherapy within 21 days before the first dose of study drug; received anti-cancer treatment other than chemotherapy or study drug treatment within 28 days (or 5 times the half-life, whichever is shorter); or have not recovered from acute toxicity related to previous treatment.

Participants with proteinuria greater than 1+ in urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria. Screeners with urine protein ≥1 g/24 hours will be ineligible for the study.

Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other conditions that may affect the absorption of lenvatinib.

Clinically symptomatic central nervous system metastases and/or carcinomatous meningitis, or a history of leptomeningeal carcinomatosis; Any other active malignant tumors within the past 24 months, except for recurrent hepatoblastoma that is the reason for participation in this study; A history of congenital or acquired immunodeficiency; Previous allogeneic stem cell or solid organ transplantation; Previous receipt of immune checkpoint inhibitors (including but not limited to pembrolizumab, nivolumab), lenvatinib, or irinotecan; A history of (non-infectious) pneumonia requiring steroid treatment or current pneumonia.

Patients with known or suspected allergic history to putilizumab or similar drugs, a history of hypersensitivity to chimeric or humanized antibodies or fusion proteins, or allergies to excipients of the study drug; A history of gastrointestinal bleeding within 4 weeks before enrollment, or a clear tendency for gastrointestinal bleeding (e.g., known active local ulcer lesions, fecal occult blood ≥++, and if persistent fecal occult blood +, gastroscopy should be performed), or other conditions judged by the investigator that may cause gastrointestinal bleeding (e.g., severe gastric fundus/esophageal varices); Cardiac diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within the past 6 months; congestive heart failure (New York Heart Association [NYHA] class >2); arrhythmias that are poorly controlled or require pacemaker treatment; hypertension uncontrolled by drugs (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);

Active infections, including:

1. Positive for human immunodeficiency virus (HIV) (HIV1/2 antibodies);
2. Active tuberculosis;
3. Other uncontrolled active infections (CTCAE V5.0 >Grade 2); Failure to recover from surgery, such as unhealed incisions or severe postoperative complications; Vaccination with any live-attenuated vaccine within 4 weeks before enrollment or likely to be administered during the study period; seasonal influenza vaccines without live viruses are allowed.

Pregnant or lactating women; A history of alcohol, psychotropic drug, or other substance abuse within the past 6 months; Any other conditions that the investigator deems make the patient ineligible for enrollment.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-04-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
PFS | PFS is defined as the time interval from the start of treatment until the occurrence of disease progression or death of the patient from any cause, whichever happens first (up to 24 months）.
  progression of the disease or the death

SECONDARY OUTCOMES:
OS | The assessment of OS will be carried out over an estimated period of up to 24 months.
  Overall survival (OS) is defined as the time from the initiation of treatment with pucotenlimab in combination with theLenvatinib and Irinotecan regimen until the patient's death from any cause. Death is determined based on official medical records or other reliable documentation. The follow - up for OS will continue throughout this estimated assessment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Yizhuo Zhang, Guangdong, Guangzhou, China